CLINICAL TRIAL: NCT01049776
Title: A Phase II Study of GW786034 in Patients With Non Small Cell Lung Cancer Who Have Failed at Least Two Prior Chemotherapy Regimens. An Institutional Pilot Study
Brief Title: GW786034 in Patients With Non Small Cell Lung Cancer 3rd Line
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated due to positive results seen in statistical analysis. Adequate patient enrollment was achieved.
Sponsor: Illinois CancerCare, P.C. (Other)
Responsible Party: Principal Investigator, Sachdev Thomas, Principal Investigator, Illinois CancerCare, P.C.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ILCC #2 IllinoisCancerCare #2
Record Dates: First submitted 2010-01-12; First posted 2010-01-14 (Estimated); Results first posted 2014-09-19 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Lung Cancer Non Small Cell
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pazapanib (GW786034) (Experimental)
  Interventions: Drug: Pazopanib (GW786034)

INTERVENTIONS:
Drug: Pazopanib (GW786034) — Pazopanib 800 mg daily x 12 weeks, (Cycle = 21 days) up to 24 months
  Other Names: Pazopanib monohydrochloride salt GW786034

SUMMARY:
Lung Cancer is the most common cause of cancer death in the United States with an estimated mortality in excess of 160,000, more than the combined mortality seen with prostate, breast, colorectal cancers(1). Most patients with Lung Cancer have Non-Small Cell Lung Cancers( NSCLC) and only 25-30% of patients with NSCLC (Non Small Cell Lung Cancer) have resectable disease( Stage I or II) at the time of diagnosis.

The vast majority of patients with advanced NSCLC (Non Small Cell Lung Cancer) are not curable and overall five year survival is 11%-14%1.

Chemotherapy is beneficial for patients with locally advanced and metastatic disease. Numerous phase III studies have determined the superiority of systemic chemotherapy over best supportive care. Platinum based chemotherapy has been widely accepted as the standard of care for the initial treatment of advanced NSCLC.

However first line chemotherapy is modest at best. A randomized trial comparing four of the most commonly used chemotherapy regimens in the United States not only failed to show a clearly superior arm but also confirmed the dismal prognosis of these patients. The response rate for all 1207 patients was 18.6% with a median survival of eight months and one year survival of 33.5 % and a two year survival of 12%5. Clearly a different paradigm is needed for the treatment of this disease.

DETAILED DESCRIPTION:
Better therapies for patients with NSCLC (Non Small Cell Lung Cancer) who progress after initial chemotherapy is urgently needed.

Besides VEGF (vascular endothelial growth factor), human lung cancers are known to express PDGFR (platelet-derived growth factor receptors). NSCLC, like most cancers, involves defects in signal transduction pathways. Receptor tyrosine kinases (RTKs) play a pivotal role in these signaling pathways, transmitting extracellular molecular signals into the cytoplasm and/or nucleus of a cell. Among such RTKs are the receptors for polypeptide growth factors such as epidermal growth factor (EGF), insulin, platelet-derived growth factor (PDGF), neurotrophins (i.e., NGF), and fibroblast growth factor (FGF). Phosphorylation of such RTKs activates their cytoplasmic domain kinase function, which in turns activates downstream signaling molecules. Thus, RTKs are key mediators of cellular signaling as well as oncogenesis resulting from over-expression and activation of such RTKs and their substrates. Due to their pivotal role in normal and aberrant signaling, RTKs are the subject of increasing focus as potential drug targets for the treatment of certain types of cancer. For example, Herceptin.RTM., an inhibitor of HER2/neu, is currently an approved therapy for a certain subset of breast cancer. Iressa.TM. (ZD1839) and Tarceva.TM. (OSI-774), both small-molecule inhibitors of EGFR, have been approved for the treatment of NSCLC.

Platelet-derived growth factor (PDGF) and its receptors (PDGFRs) are a family of RTKs that play an important role in the regulation of normal cell growth and differentiation. PDGFRs are involved in a variety of pathological processes, including atherosclerosis, neoplasia, tissue repair, and inflammation. PDGFRs, which consist of two isoforms (alpha and beta), are membrane protein-tyrosine kinases that, upon binding to PDGF, become activated and, via recruitment of SH domain-containing effector molecules, initiate distinct or overlapping signaling cascades that coordinate cellular responses.

Expression of a constitutively active PDGFR leads to cellular transformation and suggests that, in normal cells, PDGFR activity must be tightly regulated to oppose continuous activation of its downstream effectors. PDGFR beta, for example, is known to be over-expressed in a large number of tumors, and PDGF treatment causes transformation and malignant tumors in a variety of experimental systems. One study reported the apparent expression of PDGFR alpha in nearly 100% of human lung cancer tumors examined, and reported the growth inhibition of a lung cancer cell line, A549, by Gleevec, an effect that was surmised to be mediated via PDGFR inhibition.

Donnem et al evaluated 335 resected patients with stage I to III with NSCLC. Using IHC (immunohistochemical staining) the expression of PDGF-A, -B, -C and -D along with PDGFR alpha and beta. In multivariant analysis high tumor cell expression of PDGF-B and PDGF- alpha were independent negative prognostic predictors. They suggested that PDGF inhibition may be an option for treatment of NSCLC.

Socinski et al recently described the activity of sunitnib malate (SU11248) an oral, multitargeted tyrosine kinase inhibitor targeting VEGFR, PDGFR, KIT, FLT3 and RET on tumor cells, tumor neovasculature and pericytes. In an open-label, two-stage, multicenter phase II trial evaluating the single-agent activity of sunitinib in refractory NSCLC, patients with confirmed diagnosis of NSCLC, ECOG PS 0-1, no recent gross hemoptysis, no brain metastases, patients (pts) previously treated with 1-2 chemotherapy regimens, and adequate end-organ function, pts received sunitinib at 50 mg/day po for 4 weeks (wks) followed by 2 wks off treatment (6 wks considered a cycle). A total of 64 pts were enrolled and 63 pts treated. Six confirmed partial responses have been observed among 63 treated patients. Stable disease has been observed in an additional 12 pts (19.0% of all treated patients). Based on this study, Sunitinib appeared to have single-agent activity in previously treated pts with recurrent and advanced NSCLC, with the level of activity similar to currently approved agents. Sunitinib was well tolerated in this population. The trial was extended to explore a continuous dosing strategy of sunitinib at 37.5 mg/day po.

In addition to VEGF and PDGFR, expression of c-kit has been described in NSCLC. Moreover, it has been found to have an effect on survival. Micke et al, stained the tumor tissue of 95 consecutive patients with adenocarcinoma of the lung, using a polyclonal c-kit antibody. c-kit expression was correlated with relevant clinical parameters obtained by chart review. Positive c-kit expression in tumor tissue was observed in 61 of 95 patients (64%). Univariate analysis showed a significant effect of T (p = 0.003), N (p = 0.001) and M stage (p < 0.001) as well as of performance status (p = 0.001), surgical resection (p < 0.001), and LDH serum levels (p = 0.016) on survival. In contrast, c-kit protein expression was non- significant (p = 0.913). However, multivariate Cox regression with the influential parameters revealed a significant effect of c-kit expression on survival. They concluded that, the receptor tyrosine kinase c-kit is frequently expressed in adenocarcinomas of the lung and has a relevant effect on patient survival. They also concluded that the results of this study support clinical trials targeting the c-kit receptor with specific c-kit inhibitors.

Combined blockade of VEGF, PDGFR and c-kit may result in better outcomes for patients with Non Small Cell Lung Carcinoma.

Pazopanib is a novel, orally active small molecule inhibitor targeting multiple tyrosine kinases including VEGFR-1, VEGFR-2, VEGFR-3, PDGFR-alpha and - beta, and c-kit. An antitumor effect due to inhibiting of the VEGF driven angiogenic pathway is well established. In addition to its effects on VEGF receptors, pazopanib targets additional tyrosine kinases including PDGF receptors and c-kit that have established roles in tumorigenesis and oncogenic mutations in both have been described. Preliminary data from a phase I study of pazopanib in patients with solid tumors demonstrated early evidence of antitumor activity. Among 43 patients enrolled, a minimal response occurred in 4 patients and stable disease >6 months, was observed in an additional 6 patients.

Pazopanib was well tolerated at doses up to 2000 mg daily. Pazopanib is a potent and selective, orally available, small molecule inhibitor of VEGFR-1, -2, and -3, PDGF-α, PDGF-β, and c-kit tyrosine kinases (TKs). The agent selectively inhibits proliferation of endothelial cells stimulated with VEGF but not with basic fibroblast growth factor. In non-clinical angiogenesis models, pazopanib inhibited VEGF-dependent angiogenesis in a dose-dependent manner and in xenograft tumor models, twice-daily administration of pazopanib significantly inhibited tumor growth in mice implanted with various human tumor cells. Upon chronic oral dosing, pazopanib is expected to inhibit VEGF driven angiogenesis and as a consequence, limit solid tumor growth. Because angiogenesis is necessary for the growth and metastasis of solid tumors, and VEGF is believed to have a pivotal role in this process, pazopanib treatment may have broad-spectrum clinical utility.

Based on its ability to target multiple tyrosine kinases including VEGFR-1, VEGFR-2, VEGFR-3, PDGFR-alpha and beta and c-kit, which have been implicated in non small cancer, investigation of Pazopanib in patients with non small cell lung cancer is warranted.

ELIGIBILITY:
Inclusion Criteria:

Required Characteristics 3.1. Subjects must provide written informed consent prior to performance of study-specific procedures or assessments, and must be willing to comply with treatment and follow up. Procedures conducted as part of the subject's routine clinical management (e.g., blood count, imaging study) and obtained prior to signing of informed consent may be utilized for screening or baseline purposes provided these procedures are conducted as specified in the protocol.

Note: It is not necessary that informed consent be obtained within the protocol-specified screening window.

3.11 ≥18 years of age.

3.12 ≥2 prior systemic therapies for Non Small Cell Lung Cancer.

3.13 Histologic or cytologic diagnosis of stage IV Non Small Cell Lung cancer

. 3.14 Measurable disease. For patients having only lesions measuring ≥1 cm to ≤2 cm per RECIST criteria must use spiral CT imaging for both pre- and post-treatment tumor assessments.

3.15 Laboratory values obtained ≤14 days prior to registration: Hematologic Absolute neutrophil count (ANC) 1.5 X 109/L Hemoglobin1 9 g/dL (5.6 mmol/L) Platelets 100 X 109/L Prothrombin time (PT) or international normalized ratio (INR) 1.2 X upper limit of normal (ULN) Partial thromboplastin time (PTT) 1.2 X ULN Hepatic2 Total bilirubin 1.5 X ULN AST and ALT 2.5 X ULN Renal Serum creatinine 1.5 mg/dL (133 µmol/L)

Or, if greater than 1.5 mg/dL:

Calculated creatinine clearance 50 mL/min

Urine Protein to Creatinine Ratio (UPC)3 < 1

1. Subjects may not have had a transfusion within 7 days of screening assessment.
2. Concomitant elevations in bilirubin and AST/ALT above 1.0 x ULN are not permitted
3. If UPC >/= 1, then a 24-hour urine protein must be assessed. Subjects must have a 24-hour urine protein value <1g to be eligible.

   3.16 ECOG Performance Score 0, or 1.

   3.17 Negative pregnancy test done ≤ 7 days prior to registration, for women of childbearing potential only.

   A female is eligible to enter and participate in this study if she is of: Non-childbearing potential (i.e., physiologically incapable of becoming pregnant), including any female who has had:
   * A hysterectomy
   * A bilateral oophorectomy (ovariectomy)
   * A bilateral tubal ligation
   * Is post-menopausal

   Subjects not using hormone replacement therapy (HRT) must have experienced total cessation of menses for ≥ 1 year and be greater than 45 years in age, OR, in questionable cases, have a follicle stimulating hormone (FSH) value >40 mIU/mL and an estradiol value < 40pg/mL (<140 pmol/L).

   Subjects using HRT must have experienced total cessation of menses for >= 1 year and be greater than 45 years of age OR have had documented evidence of menopause based on FSH and estradiol concentrations prior to initiation of HRT

   Childbearing potential, including any female who has had a negative serum pregnancy test within 1 week prior to the first dose of study treatment, preferably as close to the first dose as possible, and agrees to use adequate contraception. GSK acceptable contraceptive methods, when used consistently and in accordance with both the product label and the instructions of the physician, are as follow:
   * An intrauterine device with a documented failure rate of less than 1% per year.
   * Vasectomized partner who is sterile prior to the female subject's entry and is the sole sexual partner for that female.
   * Complete abstinence from sexual intercourse for 14 days before exposure to investigational product, through the dosing period, and for at least 21 days after the last dose of investigational product.
   * Double-barrier contraception (condom with spermicidal jelly, foam suppository, or film; diaphragm with spermicide; or male condom and diaphragm with spermicide).
   * Oral contraceptives
   * Female subjects who are lactating should discontinue nursing prior to the first dose of study drug and should refrain from nursing throughout the treatment period and for 14 days following the last dose of study drug

   3.18 Ability and willingness to provide informed consent.

   3.19 Life expectancy ≥12 weeks.

   -

   Exclusion Criteria:

   3.21 Any of the following as this regimen may be harmful to a developing fetus or nursing child.

   • Pregnant women
   * Nursing women
   * Men or women of childbearing potential or their sexual partners who are unwilling to employ adequate contraception.

   3.22 Any abnormal serum calcium, magnesium, and potassium levels

   3.23 Clinically significant hemoptysis, cerebral hemorrhage, or gastrointestinal hemorrhage in the past 6 months

   3.24 Any patient currently on an antiarrhythmics or other medications that are know to prolong the QT interval.

   3.25 Uncontrolled infection.

   3.26 Poorly controlled hypertension [defined as systolic blood pressure (SBP) of ≥140 mmHg or diastolic blood pressure (DBP) of ≥ 90mmHg].

   Note: Initiation or adjustment of antihypertensive medication(s) is permitted prior to study entry. BP must be re-assessed on two occasions that are separated by a minimum of 1 hour; on each of these occasions, the mean (of 3 readings) SBP / DBP values from each BP assessment must be <140/90 mmHg in order for a subject to be eligible for the study

   3.27 Any condition (e.g., gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation, prior surgical procedures, affecting absorption, or active peptic ulcer disease) that impairs their ability to swallow and retain pazopanib tablets.
   * Malabsorption syndrome
   * Major resection of the stomach or small bowel. 3.28 Clinically significant gastrointestinal abnormalities that may increase the risk for gastrointestinal bleeding including, but not limited to:
   * Active peptic ulcer disease
   * Known intraluminal metastatic lesion/s with risk of bleeding
   * Inflammatory bowel disease (e.g. ulcerative colitis, Crohn's disease), or other gastrointestinal conditions with increased risk of perforation
   * History of abdominal fistula, gastrointestinal perforation, or intra abdominal abscess within 28 days prior to beginning study treatment.

   3.29 Known endobronchial lesions and or lesions infiltrating major pulmonary vessels.

   3.30 Cavitary lesions deemed to be at increased risk of bleeding.

   3.31 Any other severe underlying diseases that are, in the judgment of the investigator, inappropriate for entry into this study.

   3.32 Second primary malignancy except for carcinoma in situ of the cervix or nonmelanomatous skin cancer, unless that prior malignancy was diagnosed and definitively treated ≥5 years previously with no subsequent evidence of recurrence. Patients with a history of low-grade (Gleason score ≤6) localized prostate cancer will be eligible even if diagnosed <5 years prior to registration.

   3.33 Any ancillary therapy considered investigational (utilized for a non-FDA approved indication and in the context of a research investigation) ≤4 weeks prior to registration.

   3.34 Other concurrent chemotherapy, immunotherapy, radiotherapy.

   3.35a. History of allergic reactions attributed to compounds of similar chemical or biologic composition to pazopanib or other agents used in the study.

   b. Medications that act through the CYP450 system. Some medications that act through the cytochrome P450 system are specifically prohibited in patients receiving pazopanib. Certain other agents should be used with caution. (A list of medications that are specifically prohibited or that should be used with caution during this trial of pazopanib will be provided with the full study protocol as Appendix 1. A list of selected agents that could affect pazopanib will be listed in Appendix I. ) c. Any of the following concurrent severe and/or uncontrolled medical conditions:

   • Serious or non-healing wound, ulcer, or bone fracture

   • History of abdominal fistula, diverticulosis, gastrointestinal perforation, or intra-abdominal abscess ≤28 days prior to registration
   * Any history of cerebrovascular accident (CVA) ≤6 months prior to registration
   * History of any one or more of the following cardiovascular conditions within the past 6 months:
   * Cardiac angioplasty or stenting
   * Myocardial infarction
   * Unstable angina
   * Coronary artery bypass graft surgery
   * Symptomatic peripheral vascular disease
   * Class III or IV congestive heart failure, as defined by the New York Heart Association (NYHA)
   * History of venous thrombosis ≤12 weeks prior to registration.
   * Class III or IV heart failure as defined by the NYHA functional classification system .History of Class II heart failure and is asymptomatic on treatment may be considered eligible.
   * Poorly controlled diabetes.
   * Interstitial pneumonia or extensive and symptomatic interstitial fibrosis of the lung.
   * QTc prolongation (defined as a QTc interval ) > 480 msecs using Bazett's formula) or other significant ECG abnormalities d. Symptomatic, untreated, or uncontrolled CNS metastases or seizure disorder. Patients with CNS metastases treated with whole brain radiation (WBRT)or gamma knife may be enrolled after completion of WBRT or gamma knife. Patients may begin chemotherapy as early as the next day after completion of WBRT or gamma knife.

     e. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection or psychiatric illness/social situations that would limit compliance with study requirements.

     f. HIV-positive patients on combination antiretroviral therapy because of the potential for pharmacokinetic interactions with pazopanib. In addition, these patients are at increased risk of lethal infections when treated with marrow suppressive therapy

     g. Any of the following prior therapies:
   * Major surgery (i.e., laparotomy), open biopsy, or significant traumatic injury ≤4 weeks prior to registration. Minor surgery ≤4 weeks prior to registration. Insertion of a vascular access device is not considered major or minor surgery in this regard.
   * Treatment with any of the following anti-cancer therapies:
   * radiation therapy, surgery or tumor embolization within 14 days prior to the first dose of Pazopanib OR
   * chemotherapy, immunotherapy, biologic therapy, investigational therapy or hormonal therapy within 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of pazopanib

   Patients with progressive disease inside of the radiation field are not eligible.

   3.36 History of cerebrovascular accident including transient ischemic attack (TIA), pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months.

   Note: Subjects with recent DVT who have been treated with therapeutic anti-coagulating agents for at least 6 weeks are eligible

   3.37 Evidence of active bleeding or bleeding diathesis.

   3.38 Hemoptysis within 6 weeks of first dose of study drug.

   3.39 Unable or unwilling to discontinue use of prohibited medications for at least 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of study drug and for the duration of the study.

   3.40 Any ongoing toxicity from prior anti-cancer therapy that is >Grade 1 and/or that is progressing in severity, except alopecia.

   3.41 Other Eligibility Criteria Considerations To assess any potential impact on subject eligibility with regard to safety, the investigator must refer to the following document(s) for detailed information regarding warnings, precautions, contraindications, adverse events, and other significant data pertaining to the investigational product(s) being used in this study: Clinical Investigator's Brochure for pazopanib.[Investigator Brochure]

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-01; Primary Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sachdev P. Thomas, M.D., Principal Investigator — Illinois CancerCare, P.C.
Locations (13):
- United States (13):
  - Illinois CancerCare, P.C., Bloomington, Illinois
  - Illinois CancerCare, P.C., Canton, Illinois
  - Illinois CancerCare, P.C., Carthage, Illinois
  - Illinois CancerCare, P.C., Eureka, Illinois
  - Illinois CancerCare, P.C., Galesburg, Illinois
  - Illinois CancerCare, P.C., Macomb, Illinois
  - Illinois CancerCare, P.C., Monmouth, Illinois
  - Illinois CancerCare, P.C., Normal, Illinois
  - Illinois CancerCare, P.C., Ottawa, Illinois
  - Illinois CancerCare, P.C., Pekin, Illinois
  - Illinois CancerCare, P.C., Peoria, Illinois
  - Illinois CancerCare, P.C., Peru, Illinois
  - Illinois CancerCare, P.C., Princeton, Illinois

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pazapanib (GW786034)
Started | 32
Completed | 12
Not Completed | 20

BASELINE CHARACTERISTICS:
Population: Stratification was performed based on histology of disease. Enrollment was targeted to 21 patients with squamous histology and 21 patients with non- squamous histology. Due to the lack of patients with squamous histology, the study was closed prior to meeting the enrollment goal of 44 subjects.
Arm/Group | Pazapanib (GW786034)
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 31
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 32

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Non Small Cell Lung Cancer Participants With Disease Control (Complete Response+Partial Response+Stable Disease) Based on RECIST 1.0 Measured by CT or MRI
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions assessed by MRI or CT: Complete Response (CR), Disappearance of all target lesions: Partial Response (PR), >= 30% decrease in the sum of the longest diameter of target lesion, taking as reference the baseline sum of the longest diameter: Stable Disease (SD), Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for Progressive Disease, taking as reference the smallest sum Longest Diameter since the treatment started
Time Frame: 12 weeks
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Pazapanib (GW786034)
Number analyzed (Participants) | 32
Proportion of participants | 0.38 [0.21 to 0.56]

2. Secondary Outcome: To Describe the Clinical Toxicity Profile of Pazopanib in This Particular Patient Population
Time Frame: after the first 6 patients and quarterly
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Pazapanib (GW786034)
Serious Adverse Events (participants affected / at risk) | 11/32
Other Adverse Events (participants affected / at risk) | 32/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pazapanib (GW786034) (N=32)
Death (General disorders) | 6
Mucositis oral (Gastrointestinal disorders) | 1
Cardiac disorders - Other, specify (Cardiac disorders) | 1 — nonspecific T-wave abnormality
Upper respiratory infection (Infections and infestations) | 2
Ileus (Gastrointestinal disorders) | 1
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 — lymphopenia
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pazapanib (GW786034) (N=32)
Allergic Rhinitis (Immune system disorders) | 6
Blood/Bone Marrow- AML (Blood and lymphatic system disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 22
Leukocytes (Blood and lymphatic system disorders) | 11
Lymphopenia (Blood and lymphatic system disorders) | 25
Neutrophils (Blood and lymphatic system disorders) | 5
Platelets (Blood and lymphatic system disorders) | 19
Cardiac Arrythmia- Systolic Anterior Motion (Cardiac disorders) | 1
Cardiac Troponin I (Cardiac disorders) | 3
Hypertension (Cardiac disorders) | 22
Hypotension (Cardiac disorders) | 5
Left Ventricular Systolic Dysfunction (LVSD) (Cardiac disorders) | 1
Mitral Regurgitation (Cardiac disorders) | 1
Prolonged QTc Interval (Cardiac disorders) | 4
Supraventricular and Nodal Arrhthymia- Atrial Fibrillation (Cardiac disorders) | 2
Supraventricular and Nodal Arrhthymia- Sinus Bradycardia (Cardiac disorders) | 5
Supraventricular and Nodal Arrhthymia- Sinus Tachycardi (Cardiac disorders) | 3
Ventricular Arrythmia- PVCs (Cardiac disorders) | 1
INR (Blood and lymphatic system disorders) | 4
PTT (Blood and lymphatic system disorders) | 3
Fatigue (General disorders) | 32
Fever (Infections and infestations) | 3
Insomnia (General disorders) | 6
Rigors/Chills (General disorders) | 6
Sweating (General disorders) | 3
Weight Loss (General disorders) | 14
Dry Skin (Skin and subcutaneous tissue disorders) | 4
Hypopigmentation (Skin and subcutaneous tissue disorders) | 1
Pruritis (Skin and subcutaneous tissue disorders) | 3
Rash/desquamation (Skin and subcutaneous tissue disorders) | 12
Nail Changes (Skin and subcutaneous tissue disorders) | 1
Hot Flashes/Flushes (Endocrine disorders) | 1
Thyroid Function, low (Endocrine disorders) | 9
Thyroid Function, high (Endocrine disorders) | 2
Anorexia (Gastrointestinal disorders) | 16
Colitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 12
Dehydration (Gastrointestinal disorders) | 8
Diarrhea (Gastrointestinal disorders) | 24
Dry Mouth/Salivary Gland (Gastrointestinal disorders) | 4
Dysphagia (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 2
Heartburn/Dyspepsia (Gastrointestinal disorders) | 4
Mucositis (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 25
Taste Alteration (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 15
Esophagitis (Gastrointestinal disorders) | 1
Distention/Bloating- Abdominal (Gastrointestinal disorders) | 1
Hemorrhage, GI- Lower GI NOS (Gastrointestinal disorders) | 2
Hemorrhage, GU- Urinary NOS (General disorders) | 4
Hemorrhage, Pulmonary/Upper Respiratory- Nose (General disorders) | 4
Hemorrhage, Pulmonary/Upper Respiratory- Respiratory Tract NOS (Respiratory, thoracic and mediastinal disorders) | 2
Liver Dysfunction/Failure (Hepatobiliary disorders) | 4
Infection- Blood (Hepatobiliary disorders) | 2
Infection- Bronchitis (Hepatobiliary disorders) | 3
Infection- Lung (Pneumonia) (Hepatobiliary disorders) | 4
Infection- Respiratory Tract NOS (Hepatobiliary disorders) | 2
Infection- Sinus (Hepatobiliary disorders) | 3
Infection- Skin (Hepatobiliary disorders) | 1
Infection- Stomach (Hepatobiliary disorders) | 1
Infection- Thrush (Hepatobiliary disorders) | 3
Infection- Wound (Hepatobiliary disorders) | 1
Infection- Upper Respiratory (Hepatobiliary disorders) | 2
Infection- Urinary Tract (Hepatobiliary disorders) | 5
Infection- Upper Airway NOS (Hepatobiliary disorders) | 1
Infection- Oral Cavity (Hepatobiliary disorders) | 1
Edema: Limb (Blood and lymphatic system disorders) | 5
Albumin, serum- low (Blood and lymphatic system disorders) | 18
Alkaline Phosphatase (Blood and lymphatic system disorders) | 14
ALT (SGPT) (Blood and lymphatic system disorders) | 12
AST (SGOT) (Blood and lymphatic system disorders) | 19
Bilirubin (Blood and lymphatic system disorders) | 12
Calcium, serum- high (Blood and lymphatic system disorders) | 1
Calcium, serum- low (Blood and lymphatic system disorders) | 15
Creatinine (Blood and lymphatic system disorders) | 9
Glomerular Filtration Rate (Blood and lymphatic system disorders) | 6
Glucose, serum- high (Blood and lymphatic system disorders) | 17
Glucose, serum- low (Blood and lymphatic system disorders) | 4
Lipase (Blood and lymphatic system disorders) | 1
Magnesium, serum- high (Blood and lymphatic system disorders) | 2
Magnesium, serum- low (Blood and lymphatic system disorders) | 9
Phosphate, serum- low (Blood and lymphatic system disorders) | 5
Potassium, serum- high (Blood and lymphatic system disorders) | 7
Potassium, serum- low (Blood and lymphatic system disorders) | 10
Proteinuria (Blood and lymphatic system disorders) | 16
Sodium, serum- high (Blood and lymphatic system disorders) | 2
Sodium, serum- low (Blood and lymphatic system disorders) | 22
Triglyceride, serum- high (Blood and lymphatic system disorders) | 2
Bicarbonate, serum low (Blood and lymphatic system disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Muscle Weakness- generalized (Musculoskeletal and connective tissue disorders) | 8
Muscle Weakness- upper extremity (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal/Soft Tissue- Leg Cramps (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal/Soft Tissue- Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal/Soft Tissue- Plantar Fasciitis (Musculoskeletal and connective tissue disorders) | 1
Ataxia (Nervous system disorders) | 1
Confusion (Nervous system disorders) | 5
Dizziness (Nervous system disorders) | 10
Laryngeal Nerve Dysfunction (Nervous system disorders) | 1
Mood Alteration- Anxiety (Nervous system disorders) | 4
Neurology- Tremors (Nervous system disorders) | 2
Neuropathy: Motor (Nervous system disorders) | 4
Neuropathy: Sensory (Nervous system disorders) | 16
Seizure (Nervous system disorders) | 1
Syncope (Fainting) (Nervous system disorders) | 1
Mood Alteration- Depression (Nervous system disorders) | 2
Somnolence/Depressed Level of Consciousness (Nervous system disorders) | 1
Apnea (Nervous system disorders) | 1
Vision- Blurred Vision (Eye disorders) | 6
Vision- Diplopia (Eye disorders) | 1
Vision- Flashing Lights/Floaters (Eye disorders) | 1
Watery Eyes (Eye disorders) | 4
Pain- Abdomen (General disorders) | 13
Pain- Back (General disorders) | 13
Pain- Bone (General disorders) | 3
Pain- Chest (General disorders) | 8
Pain- External Ear (General disorders) | 1
Pain- Extremity, Limb (General disorders) | 7
Pain- Finger (General disorders) | 1
Pain- Headache (General disorders) | 10
Pain- Joint (General disorders) | 9
Pain- Muscle (General disorders) | 7
Pain- Neck (General disorders) | 2
Pain- Throat (General disorders) | 1
Pain- General NOS (General disorders) | 3
Pain- Shoulder (General disorders) | 2
Bronchospasm/Wheezing (Respiratory, thoracic and mediastinal disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 13
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 18
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 6
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2
Voice Changes/Dysathria (Respiratory, thoracic and mediastinal disorders) | 2
Hiccoughs (Hiccups/Singultus) (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis/Pulmonary Infiltrates (Respiratory, thoracic and mediastinal disorders) | 1
Cystitis (Renal and urinary disorders) | 2
Incontinence, Urinary (Renal and urinary disorders) | 1
Renal Failure (Renal and urinary disorders) | 1
Urinary Retention (Renal and urinary disorders) | 2
Urinary Frequency/Urgency (Renal and urinary disorders) | 2
Syndromes- Systemic Inflammatory Response System (SIRS) (General disorders) | 2

LIMITATIONS AND CAVEATS:
Due to the lack of patients with squamous histology, the study was closed prior to meeting the enrollment goal of 44 subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes